CLINICAL TRIAL: NCT00989157
Title: A Preliminary Comparison of the Effect of Roux-en-Y Bariatric Surgery on Blood Levels of Duloxetine
Brief Title: Effects of Gastric Bypass on Blood Levels of Duloxetine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Collaborators: University of North Dakota (Other); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, James Roerig, James L Roerig, PharmD, BCPP, Neuropsychiatric Research Institute and University of North Dakota, Neuropsychiatric Research Institute, Fargo, North Dakota
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: F1J-US-X054
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Bariatric Surgery
Keywords: Gastric Bypass; Duloxetine; Cymbalta; Pharmacokinetics
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active drug (Experimental): All subjects received drug. Single arm.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Single dose of 60 mg of duloxetine
  Other Names: Cymbalta

SUMMARY:
This study aims to determine the difference, if any, in the pharmacokinetics of duloxetine between patients who are nine to fifteen months post Roux-en-Y Bariatric Surgery and control subjects matched for body mass index (BMI), age and gender.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 and 60 years.
* Subjects must be of good general health by history and physical exam.
* Ten experimental subjects 9 to 15 months post bariatric surgery (Roux-en-Y procedure), no BMI requirement.
* Ten normal control subjects who have met the inclusion criteria and have not received bariatric surgery and who are matched to the surgery subjects according to body mass index, age and sex.
* Women of child bearing potential must be practicing an accepted method of birth control (barrier method or oral contraceptive) and have a negative pregnancy test at baseline.
* No contraindications to receiving a single capsule of 60 mg of duloxetine

Exclusion Criteria:

* Allergy to duloxetine or any of its constituents.
* Candidates who are pregnant or nursing
* Candidates currently receiving any antidepressant.
* Candidates that are determined to be poor metabolizers for CYP2D6
* Subjects who smoke or use any nicotine products
* Candidates currently receiving a medication that interacts with duloxetine.
* Candidates experiencing clinically significant, unstable neurological, hepatic, renal or cardiovascular disease.
* Candidates experiencing or with a history of vomiting or diarrhea associated with bariatric surgery
* Candidates currently or with a past history of meeting DSM-IV diagnostic criteria for schizophrenia, schizoaffective disorder, bipolar disorder.
* Candidates who have participated in an investigational drug study in past 30 days.
* Candidates who meet DSM-IV diagnostic criteria for drug/alcohol abuse or dependency or who have a history of drug/alcohol abuse or dependency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Roerig, PharmD, BCPP, Principal Investigator — Neuropsychiatric Research Institute and University of North Dakota
Locations (1):
- Neuropsychiatric Research Institute, Fargo, North Dakota, United States

REFERENCES:
- See also: Neuropsychiatric Research Institute — http://www.nrifargo.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Matched to bariatric subject via BMI, age and gender
- Bariatric: One year post surgery
Period: Overall Study
Arm/Group | Control | Bariatric
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Available Bariatric surgery candidates and pilot study results.
Groups:
- Bariatric: Subjects 1 year post bariatric surgery 9 to 15 months post-RYGBP
- Control: Subjects matched to the bariatric subjects via BMI, age and gender
- Total: Total of all reporting groups
Arm/Group | Bariatric | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.10 (9.02) | 45.9 (8.54) | 45 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: The difference, if any, in the pharmacokinetics parameters (Cmax) of duloxetine between patients who are nine to fifteen months post Roux-en-Y Bariatric Surgery and control subjects matched for BMI, age and gender.
Time Frame: 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.25, 2.5, 3.5, 4.5, 6.5, 8.5, 10.5, 24, 48. 72
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Bariatric | Control
Number analyzed (Participants) | 10 | 10
ng/ml | 51.04 (11.88) | 61.41 (34.93)

2. Secondary Outcome: Emesis
Description: episodes of emesis.
Time Frame: 4 days
Measure: Number; unit: number of occurences
Groups:
- Bariatric: Subjects one year post surgery
Arm/Group | Bariatric | Control
Number analyzed (Participants) | 10 | 10
number of occurences | 2 | 3

3. Primary Outcome: Tmax
Description: Time to maximum plasma concentration
Time Frame: 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.25, 2.5, 3.5, 4.5, 6.5, 8.5, 10.5, 24, 48. 72
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Bariatric | Control
Number analyzed (Participants) | 10 | 10
Hours | 2.2 (0.86) | 6 (2.17)

4. Primary Outcome: AUCo-inf,
Description: Area under the plasma concentration time curve
Time Frame: 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.25, 2.5, 3.5, 4.5, 6.5, 8.5, 10.5, 24, 48. 72
Measure: Mean (Standard Deviation); unit: ng h/mL
Arm/Group | Bariatric | Control
Number analyzed (Participants) | 10 | 10
ng h/mL | 646.74 (79.70) | 1119.91 (593.40)

5. Primary Outcome: T1/2
Description: Half life
Time Frame: 0, 0.25, 0.5, 0.75, 1.0, 1.25, 1.5, 1.75, 2.25, 2.5, 3.5, 4.5, 6.5, 8.5, 10.5, 24, 48. 72
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bariatric | Control
Number analyzed (Participants) | 10 | 10
hours | 12.0 (0.87) | 11.75 (2.38)

ADVERSE EVENTS:
Arm/Group | Bariatric | Control
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bariatric (N=10) | Control (N=10)
Emesis (Gastrointestinal disorders) | 2 (2) | 3 (3) — Emesis post drug ingestion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No